CLINICAL TRIAL: NCT00080977
Title: Treatment of Patients With Metastatic Renal Cell Carcinoma Who Have Failed Low Dose Intensity Interleukin-2 With High-Dose Intravenous Recombinant Interleukin-2
Brief Title: High-Dose Intravenous Interleukin-2 in Treating Patients With Metastatic Renal Cell Carcinoma (Kidney Cancer) That Has Not Responded to Previous Low-Dose Intravenous or Subcutaneous Interleukin-2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Blumenthal Cancer Center at Carolinas Medical Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000357581; CMC-10-01-01AH
Record Dates: First submitted 2004-04-07; First posted 2004-04-08 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2005-06

CONDITIONS: Kidney Cancer
Keywords: recurrent renal cell cancer; stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — aldesleukin

INTERVENTIONS:
Biological: aldesleukin

SUMMARY:
RATIONALE: Interleukin-2 may stimulate a person's white blood cells to kill renal cell carcinoma (kidney cancer) cells.

PURPOSE: This phase II trial is studying how well high-dose intravenous interleukin-2 works in treating patients with metastatic renal cell carcinoma that has not responded to previous low-dose intravenous or subcutaneous interleukin-2.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate (complete, partial, and minor) in patients with metastatic renal cell carcinoma who failed prior low-dose intravenous or subcutaneous interleukin-2 (IL-2) when treated with high-dose intravenous IL-2.
* Determine the overall survival, disease-free survival, and time to progression in patients treated with this drug.
* Determine the toxicity of this drug in these patients.

OUTLINE: This is a pilot study.

Patients receive high-dose interleukin-2 IV every 8 hours for 15 doses followed 7-10 days later by another 15 doses (course 1).

Patients are assesed for response 2 months after initiation of treatment. Patients with responding or stable disease receive a second course of therapy. Patients with an ongoing response receive subsequent courses of treatment in the absence of unacceptable toxicity.

Patients are followed every 6 months for survival.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed renal cell carcinoma

  * Metastatic disease
  * No pure papillary or sarcomatoid variants
* Measurable disease
* Failed prior subcutaneous OR intravenous (dose ≤ 50,000 IU/kg/day) interleukin-2

  * Documented disease progression
* No estimated hepatic replacement by tumor > 25% by CT scan or MRI
* No tumor involving the CNS or a major nerve

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 80-100%

Life expectancy

* More than 3 months

Hematopoietic

* Platelet count ≥ 80,000/mm^3
* No sites of ongoing bleeding

Hepatic

* See Disease Characteristics
* Bilirubin ≤ 1.4 mg/dL
* AST and ALT ≤ 3 times normal
* PT or PTT INR ≤ 1.2
* Hepatitis B surface antigen negative
* Hepatitis C virus negative
* No coagulation disorders

Renal

* Creatinine ≤ 1.6 mg/dL

Cardiovascular

* No ongoing ischemia*
* No cardiac dysfunction*
* No abnormal ejection fraction* NOTE: *A cardiac stress test is indicated for all patients ≥ 50 years of age and for any patient with possible cardiac disease as suggested by history, physical exam, or electrocardiogram

Pulmonary

* FEV_1 ≤ 65% of predicted*
* Vital capacity ≤ 65% of predicted* NOTE: *Pulmonary function tests are to be performed on any patient with a significant smoking history or suspected pulmonary disease either by history, physical exam, or radiograph

Other

* HIV negative
* No AIDS
* No systemic infections
* No other malignancy except carcinoma in situ
* No psychiatric illness that would preclude study participation or compliance
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics

Chemotherapy

* Not specified

Endocrine therapy

* No concurrent steroids

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* More than 28 days since other prior treatment for renal cell cancer
* No concurrent immunosuppressive agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-06

CONTACTS AND LOCATIONS:
Overall Officials: Richard L. White, MD, Study Chair — Blumenthal Cancer Center at Carolinas Medical Center
Locations (1):
- Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina, United States